CLINICAL TRIAL: NCT03397381
Title: Outcome of Arterio-venous Fistula for Adult Hemodialysis Patients in Assiut Governorate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanan Sayed Hassan Mahrous, director of Renal dialysis Unit of Assiut Health directorate, Assiut University
Other Study IDs: 17200155
Record Dates: First submitted 2017-12-26; First posted 2018-01-12 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
identification of the factors that affect the outcome of arteriovenous fistula in chronic renal failure patients that newly established regular dialysis in Assiut Governorate

1. To study the factors that influence the outcome of AVF
2. To evaluate the vascular complications of AVF as occlusion, rupture, aneurysmal dilation and hand ischemia

ELIGIBILITY:
Inclusion Criteria:

* all adult hemodialysis Patients in Assiut Government are eligible for enrollment if they are newly dialyzed via AVF and agree to participate in the study

Exclusion Criteria:

* Patients are not dialyzed with AVF

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic renal Failure on regular dialysis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
the number of new renal failure patients with failed arteriovenous fistula as measured with arteriovenous duplex ultrasound imaging peak systolic velocity and end-diastolic velocity in Assiut Governorate | 3 years
  the arteriovenous fistula will be named fail if one or more of the following
  1. No Doppler signal
  2. Ratio of peak systolic velocity at stenosis to peak systolic velocity at 2 cm beyond anastomosis (if normal)appearing >3
  3. Intraluminal echogenicity
  4. Graft walls appear collapsed

SECONDARY OUTCOMES:
the number deaths of renal failure patients on regular dialysis related to AVF complications in Assiut Governorate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hanan S Mahrous, MD, Principal Investigator — Assiut University
Locations (1):
- Hanan, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stolic R. Most important chronic complications of arteriovenous fistulas for hemodialysis. Med Princ Pract. 2013;22(3):220-8. doi: 10.1159/000343669. Epub 2012 Nov 2. PMID 23128647
- [Result] Lok CE. Fistula first initiative: advantages and pitfalls. Clin J Am Soc Nephrol. 2007 Sep;2(5):1043-53. doi: 10.2215/CJN.01080307. Epub 2007 Aug 16. No abstract available. PMID 17702726
- [Result] Valliant A, McComb K. Vascular Access Monitoring and Surveillance: An Update. Adv Chronic Kidney Dis. 2015 Nov;22(6):446-52. doi: 10.1053/j.ackd.2015.06.002. PMID 26524949
- [Result] Hammes M. Hemodynamic and biologic determinates of arteriovenous fistula outcomes in renal failure patients. Biomed Res Int. 2015;2015:171674. doi: 10.1155/2015/171674. Epub 2015 Oct 1. PMID 26495286
- [Result] Padberg FT Jr, Calligaro KD, Sidawy AN. Complications of arteriovenous hemodialysis access: recognition and management. J Vasc Surg. 2008 Nov;48(5 Suppl):55S-80S. doi: 10.1016/j.jvs.2008.08.067. PMID 19000594